CLINICAL TRIAL: NCT02297074
Title: Evaluation of Glycemic Index Glycemic Load and Insulinemic Index of Spanish Breads and Their Effect on Incretins and Gastrointestinal Hormones Related With Appetite Regulation
Brief Title: Evaluation of Glycemic Index, Glycemic Load and Insulinemic Index of Spanish Breads
Acronym: BREADGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organización Interprofesional Agroalimentaria de Cereales Panificables y Derivados (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BreadGI
Record Dates: First submitted 2014-10-31; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
Keywords: Bread; Glycemic index; Glycemic load; Insulinemic index; Satiety; Gastrointestinal hormones
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ordinary White Bread (Experimental): Ordinary white bread bread is characterised by a white crumb with regular soft alveoli and a slightly soft thin crust.
  Interventions: Other: Ordinary white bread
- Precooked-Frozen White Bread (Experimental): Precooked-Frozen white bread is characterized by white crumb with regular soft alveoli and bright crusty crust
  Interventions: Other: Precooked-Frozen White Bread
- Candeal-flour White Bread (Experimental): Candeal-flour white bread has a thick crust of between one and two millimetres, which is smooth and crisp, golden to light brown in colour and which tastes of toasted cereal. The crumb of the bread is white and its texture is smooth, spongy and consistent, with little regular alveolus and with an intense cereal aroma with a pleasant and slightly sweet taste
  Interventions: Other: Candeal-flour White Bread
- Alfacar White Bread (Experimental): Alfacar white bread is made according to its protected designation of origin and protected geographical indication (D.O. Alfacar, Granada, Spain). The bread has a creamy white, flexible and soft crumb, with many randomly scattered holes. The crust is medium-thick to thick, golden, slightly shiny and quite smooth
  Interventions: Other: Alfacar White Bread
- Organic Wholemeal Bread (Experimental): The Organic wholemeal bread only includes organic whole grain flours as the unique difference compared with the Ordinary bread. The resulting dark brown bread is characterized by compact crumb free of alveoli and hard thin crust
  Interventions: Other: Wholemeal Bread
- Glucose (Active Comparator): Glucose is used to calculate glycemic index, glycemic load and insulinemic index
  Interventions: Other: Glucose

INTERVENTIONS:
Other: Ordinary white bread — The evening before the test day, subjects consumed a standardised dinner. Volunteers arrived in a 12-h fasting state. A fasting blood sample was acquired after the resting time, and appetite feelings were assessed by using visual analogue The subjects were instructed to consume the tested bread or 50 g of glucose. The subjects immediately completed two VAS, one on appetite feelings and another on bread palatability. The appetite feeling VAS were repeated every 30 min until a total of 180 min had passed. The subjects were not allowed to eat or drink anything else during the 180 min of the intervention.
  After the last blood extraction (3 h), an ad libitum lunch and 300 ml of water was provided. Volunteers ate until comfortably satisfied and the amount of food intake was registered
  Arms: Ordinary White Bread
Other: Precooked-Frozen White Bread — The evening before the test day, subjects consumed a standardised dinner. Volunteers arrived in a 12-h fasting state. A fasting blood sample was acquired after the resting time, and appetite feelings were assessed by using visual analogue The subjects were instructed to consume the tested bread or 50 g of glucose. The subjects immediately completed two VAS, one on appetite feelings and another on bread palatability. The appetite feeling VAS were repeated every 30 min until a total of 180 min had passed. The subjects were not allowed to eat or drink anything else during the 180 min of the intervention.
  After the last blood extraction (3 h), an ad libitum lunch and 300 ml of water was provided. Volunteers ate until comfortably satisfied and the amount of food intake was registered
  Arms: Precooked-Frozen White Bread
Other: Candeal-flour White Bread — The evening before the test day, subjects consumed a standardised dinner. Volunteers arrived in a 12-h fasting state. A fasting blood sample was acquired after the resting time, and appetite feelings were assessed by using visual analogue The subjects were instructed to consume the tested bread or 50 g of glucose. The subjects immediately completed two VAS, one on appetite feelings and another on bread palatability. The appetite feeling VAS were repeated every 30 min until a total of 180 min had passed. The subjects were not allowed to eat or drink anything else during the 180 min of the intervention.
  After the last blood extraction (3 h), an ad libitum lunch and 300 ml of water was provided. Volunteers ate until comfortably satisfied and the amount of food intake was registered
  Arms: Candeal-flour White Bread
Other: Alfacar White Bread — The evening before the test day, subjects consumed a standardised dinner. Volunteers arrived in a 12-h fasting state. A fasting blood sample was acquired after the resting time, and appetite feelings were assessed by using visual analogue The subjects were instructed to consume the tested bread or 50 g of glucose. The subjects immediately completed two VAS, one on appetite feelings and another on bread palatability. The appetite feeling VAS were repeated every 30 min until a total of 180 min had passed. The subjects were not allowed to eat or drink anything else during the 180 min of the intervention.
  After the last blood extraction (3 h), an ad libitum lunch and 300 ml of water was provided. Volunteers ate until comfortably satisfied and the amount of food intake was registered
  Arms: Alfacar White Bread
Other: Wholemeal Bread — The evening before the test day, subjects consumed a standardised dinner. Volunteers arrived in a 12-h fasting state. A fasting blood sample was acquired after the resting time, and appetite feelings were assessed by using visual analogue The subjects were instructed to consume the tested bread or 50 g of glucose. The subjects immediately completed two VAS, one on appetite feelings and another on bread palatability. The appetite feeling VAS were repeated every 30 min until a total of 180 min had passed. The subjects were not allowed to eat or drink anything else during the 180 min of the intervention.
  After the last blood extraction (3 h), an ad libitum lunch and 300 ml of water was provided. Volunteers ate until comfortably satisfied and the amount of food intake was registered
  Arms: Organic Wholemeal Bread
Other: Glucose — 50 g of glucose were administered as a reference
  Arms: Glucose

SUMMARY:
The present study was carried out to determine the glycaemic index (GI), glycaemic load (GL), insulinaemic index (InI), appetite ratings and postprandial plasma concentrations of gastrointestinal hormones related to the control of food intake after the ingestion of five types of commercially available selected Spanish breads. All volunteers took the breads and glucose in a crossover interventional study.

DETAILED DESCRIPTION:
The most important cereal-derived nourishment is bread, a staple food which is the main source of daily carbohydrates. White bread is the one for which the most rapid decline has occurred, probably due to a popular belief that bread provokes weight gain, but more studies are needed to clarify the relationship between bread consumption and ponderal status in Spanish population.

A growing body of evidence supports a beneficial role for low-glycaemic index (GI) and glycaemic load (GL) diets in the prevention of life style-related diseases such as type-2 diabetes. Likewise, GI s widely used in the selection of foods suitable for glycaemic control, since low to moderate GI diets have been proposed for the prevention of type 2 diabetes, cardiovascular disease and age-related eye diseases. On the contrary, related to obesity, no associations between BMI, GI and GL have been reported in a Mediterranean population. Thus, investigations focuses on the implication of glycaemic response of different breads are of important application.

Many factors such as manufacturing bread conditions, starch structure, bread particle size and inclusion of different types of ingredients like whole-grains may influence glycaemic response and therefore may contribute to modify GI, GL and InI of breads. Comparing different French breads, GI value varied between 57 for the traditional baguette and 85 for the wholemeal loaf, while the traditional baguette exerted a significantly lowest postprandial insulin response and the lowest InI. However, to our best knowledge, neither the influence of different types of Spanish breads on GI, GL and InI nor the effects on appetite ratings and on the postprandial gastrointestinal hormone responses have been investigated.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years old
* body mass index (BMI) between 18 and 30, normal and overweight
* healthy
* Accept to participate in the study

Exclusion Criteria:

* age below 18 and more than 45 years old
* BMI lower than 18 and more than 29
* smokers
* pregnancy or breastfeeding
* unusual fibre consumption
* glucose plasma levels higher than 110 mg/dl
* insulin plasma levels higher than 10 mU/ml
* blood pressure higher than 110 mmHg
* medication to treat blood pressure glucose or lipid metabolism
* suffering from metabolic or gastrointestinal syndrome
* genetic dyslipidemia or intake nutritional supplements in the last three months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Postprandial determination of Glycemic index and glycemic load | from fasting to 180 mins after the intake of the breads
  Glycemic index is defined as the blood glucose response measured as AUC in response to a test food consumed by an individual under standard conditions related to the postprandial response to 50 g of oral glucose load under the same conditions.
  Glycemic load takes into account the GI of the product and how many available carbohydrates are in a food serving and is calculated as GL = [GI of product/100 x g of available carbohydrates in a food serving]

SECONDARY OUTCOMES:
Postprandial determination of Insulinemic index | from fasting to 180 mins after the intake of the breads
  insulinemic index measures the increment of insulin AUC over two hours in response to consumption of the amount of bread providing a 50 g of available carbohydrates divided by AUC after ingestion of 50 g of glucose after two hours
Postprandial determination of Appetite profile | from fasting to 180 mins after the intake of the breads
  Appetite profile was assessed using VAS ratings of hunger, fullness, desire to eat and prospective food consumption, based on a 100-mm scale ranging from 0 ("not at all") to 100 ("extremely"). This questionnaire was completed before and every 30 min during the 240 min following the intake of the breakfast. A validated composite appetite score was calculated using the following equation: Composite appetite score = (satiety + fullness + (l00 - prospective food consumption) + (100 - hunger))/4 (Flint et al., 2000).
Postprandial determination of Plasma gastrointestinal hormone concentrations | from fasting to 180 mins after the intake of the breads
  For the determination of gastrointestinal hormone plasma concentrations, whole blood was added to peptidase inhibitor, which are needed for the determination of some hormones. This blood sample was centrifuged at 1000 x g for 10 min at 4 ºC, divided into aliquots and frozen at -80ºC for analyses. Plasma concentrations of insulin, ghrelin, GLP-1, gastric inhibitory polypeptide (GIP), peptide YY (PYY) and pancreatic polypeptide (PP) were determined using a MILLIplexTM kit (Millipore, USA).

CONTACTS AND LOCATIONS:
Overall Officials: MARÍA D MESA, PhD, Principal Investigator — Universidad de Granada; ANGEL GIL, PROFESSOR, Study Director — Universidad de Granada

REFERENCES:
- [Result] Barclay AW, Petocz P, McMillan-Price J, Flood VM, Prvan T, Mitchell P, Brand-Miller JC. Glycemic index, glycemic load, and chronic disease risk--a meta-analysis of observational studies. Am J Clin Nutr. 2008 Mar;87(3):627-37. doi: 10.1093/ajcn/87.3.627. PMID 18326601
- [Result] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136